CLINICAL TRIAL: NCT05286723
Title: Effectiveness Multicomponent Exercise Programme in Older Subjects. A Pilot Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER202107B
Record Dates: First submitted 2022-02-25; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Old Age; Debility; Sarcopenia; Exercise Addiction
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicomponent Training (Experimental): Traditional training. 3 times a week
  Warm-up:
  Main work:
  Aerobic training Strength training Balance and coordination training Return to calm
  Interventions: Other: Multicomponent Training

INTERVENTIONS:
Other: Multicomponent Training — Warm up, aerobic training, stenght training, balance and coordination training and return to calm

SUMMARY:
Sarcopenia can occur or increase due to sedentary lifestyles, physical inactivity or chronic endocrine and inflammatory disorders, this pathology is much more frequent in older people due to the added risk factors and the fact that the physiological ageing process generates a pro-inflammatory situation and an alteration in the synthesis of hormones and myokines, it has been observed that the loss of strength causes functional deterioration and a significant increase in the person's dependence, reduces their functional status and quality of life, and may increase the risk of falls, thereby increasing mortality.

The hipotesis of this study is that multicomponent training 3 times a week for 6 weeks, produces improvements in the functional capacity of elderly patients.

This study has the objective is whether multicomponent training 3 times a week for 6 weeks produces improvements in the functional capacity of elderly patients.

The methodology is a pilot clinical trial. The study population is people over 65 years of age, sedentary, with functional independence and with a state of health that allows them to carry out physical activity. The study is planned as a pilot study and will consist of 13 subjects in the experimental group (multicomponent training).

The variables to be measured are anthropometric variables and variables of neuromuscular function an functionality.

The intervention will be a training will be 3 times a week during 6 weeks, with a warm-up, a main block with aerobic work, strength work and training and coordination work, and finally a return to calm.

DETAILED DESCRIPTION:
Sarcopenia can occur or increase due to sedentary lifestyles, physical inactivity or chronic endocrine and inflammatory disorders, this pathology is much more frequent in older people due to the added risk factors and the fact that the physiological ageing process generates a pro-inflammatory situation and an alteration in the synthesis of hormones and myokines, it has been observed that the loss of strength causes functional deterioration and a significant increase in the person's dependence, reduces their functional status and quality of life, and may increase the risk of falls, thereby increasing mortality.

The hipotesis of this study is that multicomponent training 3 times a week for 6 weeks, produces improvements in the functional capacity of elderly patients.

This study has the objective is whether multicomponent training 3 times a week for 6 weeks produces improvements in the functional capacity of elderly patients.

The methodology is a pilot clinical trial. The study population is people over 65 years of age, sedentary, with functional independence and with a state of health that allows them to carry out physical activity. The study is planned as a pilot study and will consist of 13 subjects in the experimental group (multicomponent training).

The variables to be measured are anthropometric variables and variables of neuromuscular function an functionality.

The variables to be measured are anthropometric variables such as height, sex, age, lower limb dominance and bioimpedance, we will also measure variables of neuromuscular function, with Tensiomyography: Contraction time (Tc), and radial displacement (Dm), Myotonometry: Stiffness, Surface electromyography: %RMS, all of this in muscles Rectus femoris, vastus lateralis, vastus medialis, lateral gastrocnemius and tibialis anterior. Manual dynamometry: Peak force (Kg) grip strength (Handgrip). Information on functionality with Short Physical Performance Battery (SPPB), velocity in 4 meters walking, Timed get up and go (TUG).

The intervention will be a training will be 3 times a week during 6 weeks, with a warm-up, a main block with aerobic work, strength work and training and coordination work, and finally a return to calm.

The intervention will be a training 3 times a week with, warm up, articular and functional exercises with one's own body weight, principal work: Aerobic training 20 minutes waking then strenght training 25 minutes, i.Sets: start with 1 set to consolidate the technique, and progress to 3 sets.

ii.Repetitions: start with 10-15 repetitions (at lower intensity) and progress to 8-12 repetitions.

iii.Intensity: start with a lower intensity (even 20-30%1RM) and progress to 70-80%1RM.

iv.Rest: Breaks between sets of 3-5 minutes should be taken to avoid muscle fatigue.

v.Exercises: Leg press on machine Balance and co-ordination training during 5-10 minutes finally return to calm during 5 minutes with stretching.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary persons between 65 and 95 years of age.
* Have a walking speed ≤0.8 metres per second as this is characteristic of patients with or with onset of sarcopenia.
* Have a grip strength <30 kg for men and <20 kg for women as being characteristic of patients with or with onset of sarcopenia.

Exclusion Criteria:

* Severe untreated osteoporosis.
* Having suffered a bone fracture in the last year.
* Having had juvenile osteoporosis during adolescence or young adulthood.
* Active chronic pathology
* Uncontrolled arterial hypertension.
* Uncontrolled orthostatic hypotension.
* Severe acute respiratory failure.
* Diabetes mellitus with acute decompensation or uncontrolled hypoglycaemia.
* Endocrine, haematological and other associated rheumatic diseases.
* Mental health problems (schizophrenia, dementia, depression, etc.) or not being in full mental capacity.
* Patients with pharmacological treatments of glucocorticoids, anticoagulants and/or diuretics.
* Patients with coagulation problems or previous cardiac pathology.
* People with a body mass index (BMI) of 30 or more.
* Subjects with a systemic disease or any other pathology in which therapeutic exercise may be contraindicated.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Functionality (Running speed in 4 metres. Seconds) | Change between baseline and 6 weeks
  The participant's speed in covering 4 metres at their usual walking speed is assessed. The shorter the time, the faster the walking speed and therefore the better the functionality.
Functionality (Timed get up and go. Seconds) | Change between baseline and 6 weeks
  The time it takes the participant to get up from a chair, walk 3 metres, turn around an obstacle (a cone) and sit back down in the chair is assessed. The less time the participant takes to perform the test, the better the functionality.

SECONDARY OUTCOMES:
Functionality (Short Physical Performance Battery. 0-12 points) | Change between baseline and 6 weeks
  It consists of a battery of three exercises with a maximum score of 4 points each. The first exercise assesses the participant's balance, the second exercise assesses walking speed and the third exercise assesses the strength of the lower limbs to stand up and sit down from the chair. The maximum SPPB score is 12 points indicating excellent functionality.
Neuromuscular Function, Handgrip (Kg) | Change between baseline and 6 weeks
  A hand-held dynamometer shall be used to assess the maximum grip force for 5 seconds. The participant shall squeeze the dynamometer as hard as possible and the dynamometer shall record the force applied.
Neuromuscular Function, Myotonometry (Stiffness) | Change between baseline and 6 weeks
  Myotonometry is an instrument that assesses the viscoelasticity of tissue by means of a mechanical impulse in the muscle belly. The device generates a small mechanical impulse in the muscle belly and, depending on the response of the muscle belly to this stimulus, provides the variable stiffness.
Neuromuscular Function,Tensiomyography (Radial displacement (Dm)). | Change between baseline and 6 weeks
  Tensiomyography is an instrument which, at a given power, generates an involuntary muscle contraction in the muscle under examination. The contraction causes a movement of the muscle belly in a radial direction which is detected by a mechanical sensor placed just in contact with the muscle. The mechanical sensor collects the variables of radial displacement (Dm).
Neuromuscular Function,Tensiomyography (Shrinkage time (Tc)) | Change between baseline and 6 weeks
  Tensiomyography is an instrument which, at a given power, generates an involuntary muscle contraction in the muscle under examination. The contraction causes a movement of the muscle belly in a radial direction which is detected by a mechanical sensor placed just in contact with the muscle. The mechanical sensor collects the variables of contraction time (Tc).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain